CLINICAL TRIAL: NCT06583681
Title: Shape of the Sagittal Curvatures of the Spine in Youthful Female Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Ewa Puszczalowska-Lizis, MsPT, PhD Professor (Associate), University of Rzeszow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 05072024
Record Dates: First submitted 2024-07-05; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Sport; Training; Kyphosis; Lordosis; Health
MeSH Terms: conditions — Kyphosis; Lordosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sagittal curvatures of the spine (Other): The measuring of the sagittal curvatures of the spine.
  Interventions: Other: The measuring of the sagittal curvatures of the spine

INTERVENTIONS:
Other: The measuring of the sagittal curvatures of the spine — Research tool was Baseline Bubble inclinometer.

SUMMARY:
The goal of this study is to assess the formation of the sagittal curvatures of the spine in healthy girls practicing volleyball versus their untrained peers.

Research questions:

1. Is there a differentiation in values of thoracic kyphosis, lumbar lordosis angles, and compensation ratio among girls practicing volleyball and their untrained peers?
2. Does practicing volleyball determine the frequency of correctness in the lumbosacral inclination, the shape of the curvature of the thoracic kyphosis and lumbar lordosis?
3. Does practicing volleyball determine the frequency of types and subtypes of body posture?

DETAILED DESCRIPTION:
The investigators compared 30 healthy girls aged 10-13 (attending training regularly, three times a week), with 30 healthy peers who did not train in any sports and did not regularly participate in any physical exercises apart from attending obligatory physical education classes. The Baseline Bubble inclinometer was applied as the research tool of choice. The study protocol entailed the measuring of the sagittal curvatures of the spine.

ELIGIBILITY:
Inclusion Criteria:

* age range of 10-13 years,
* dominating right hand and right leg,
* a written informed consent to participate in the study.

Exclusion Criteria:

* injuries of the musculoskeletal system,
* pathology of the limbs,
* previous orthopedic surgery,
* neurological disorders,
* refusal to participate in the study.

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced abnormalities resulting from sports training according to inclinometer assessment | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Puszczalowska-Lizis, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszow, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No